CLINICAL TRIAL: NCT07081958
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center, Phase II Study to Evaluate the Efficacy, Safety, and Tolerability of Once-Daily RO7795081 Administered for 38 Weeks to Participants With Obesity or Overweight With at Least One Weight-Related Comorbidity
Brief Title: A Study Evaluating the Effect of Daily Oral RO7795081 in Participants With Obesity or Overweight With at Least One Weight-Related Comorbidity
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP45702
Record Dates: First submitted 2025-07-22; First posted 2025-07-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Obesity or Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2: RO7795081 Dosing Regimen 1 (Experimental)
  Interventions: Drug: RO7795081
- Arm 3: RO7795081 Dosing Regimen 2 (Experimental)
  Interventions: Drug: RO7795081
- Arm 4: RO7795081 Dosing Regimen 3 (Experimental)
  Interventions: Drug: RO7795081
- Arm 5: RO7795081 Dosing Regimen 4 (Experimental)
  Interventions: Drug: RO7795081
- Arm 6: RO7795081 Dosing Regimen 5 (Experimental)
  Interventions: Drug: RO7795081
- Arm 7: RO7795081 Dosing Regimen 6 (Experimental)
  Interventions: Drug: RO7795081
- Arm 8: RO7795081 Dosing Regimen 7 (Experimental)
  Interventions: Drug: RO7795081

INTERVENTIONS:
Drug: RO7795081 — RO7795081 will be administered orally once daily, according to the randomized dosing regimen, during the 38-week treatment period.
  Other Names: CT-996; RG6652
  Arms: Arm 2: RO7795081 Dosing Regimen 1; Arm 3: RO7795081 Dosing Regimen 2; Arm 4: RO7795081 Dosing Regimen 3; Arm 5: RO7795081 Dosing Regimen 4; Arm 6: RO7795081 Dosing Regimen 5; Arm 7: RO7795081 Dosing Regimen 6; Arm 8: RO7795081 Dosing Regimen 7
Drug: Placebo — Placebo matching each RO7795081 dosing regimen arm will be administered orally once daily during the 38-week treatment period.
  Arms: Arm 1: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-range-finding, Phase II study aims to evaluate the efficacy, tolerability, and safety of RO7795081 for chronic weight management in adult participants with obesity or overweight with at least one weight-related comorbidity, but without diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have at screening:

  1. Body mass index (BMI) greater than or equal to (≥)30.0 kg/m^2; or
  2. BMI ≥27.0 kg/m^2 and <30.0 kg/m^2 with at least one weight-related comorbidity, such as hypertension, dyslipidemia, diagnosis of obstructive sleep apnea, cardiovascular disease
* History of ≥1 self-reported unsuccessful diet/exercise effort to lose body weight
* A stable body weight for the 3 months prior to screening (maximum 5% body weight gain and/or loss)

Exclusion Criteria:

* Have a history or diagnosis of any type of diabetes mellitus (Type 1 diabetes [T1D], T2D, or rare forms of diabetes)
* Have obesity induced by other endocrinologic disorders (e.g., Cushing's syndrome) or diagnosed monogenetic or syndromic forms of obesity (e.g., melanocortin-4 receptor deficiency or Prader-Willi Syndrome)
* Participation in unbalanced/extreme diets or in an organized weight reduction program within 3 months of the screening visit or planning to engage in such diets or programs during the study
* Prior or planned surgical treatment for obesity
* Have a known, clinically significant gastric emptying abnormality
* Have poorly controlled hypertension, untreated renal artery stenosis, or evidence of labile blood pressure including symptomatic postural hypotension
* Have any of the following cardiovascular conditions within 3 months prior to screening: Acute myocardial infarction; Cerebrovascular accident (stroke)/transient ischemic attack; Unstable angina; Hospitalization due to congestive heart failure.
* Have a history of acute or chronic pancreatitis
* Have a history of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder (e.g., schizophrenia, bipolar disorder, or other serious mood or anxiety disorder), or had a suicide attempt within the last 1 year of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Body Weight From Baseline to Week 30 | Baseline to Week 30

SECONDARY OUTCOMES:
Absolute Change in Body Weight (kg) from Baseline to Week 30 | Baseline to Week 30
Absolute Change in Body Weight (kg) from Baseline to Week 38 | Baseline to Week 38
Percent Change in Body Weight From Baseline to Week 38 | Baseline to Week 38
Percentage of Participants Who Achieve ≥5%, ≥10%, ≥15%, or ≥20% Body Weight Reduction from Baseline at Week 30 | Baseline and Week 30
Percentage of Participants Who Achieve ≥5%, ≥10%, ≥15%, or ≥20% Body Weight Reduction from Baseline at Week 38 | Baseline and Week 38
Absolute Change in BMI (kg/m^2) from Baseline to Week 30 | Baseline to Week 30
Absolute Change in BMI (kg/m^2) from Baseline to Week 38 | Baseline to Week 38
Incidence of Adverse Events (AEs), Adverse Events of Special Interest (AESIs), and Serious AEs (SAEs) | From first dose until 28 days after the final dose of study treatment (42 weeks)
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) Scores from Baseline to Week 42 | Baseline to Week 42
  The C-SSRS is an assessment tool to evaluate suicidal ideation and behavior during the assessment period via a participant-reported questionnaire comprising 2 to 6 questions (yes or no). Affirmative responses count as 1 point, which are then summed to indicate the level of suicide risk on a scale of 0 (no risk) to 6 (high risk).
Change in Patient Health Questionnaire-9 (PHQ-9) Scores from Baseline to Week 42 | Baseline to Week 42
  PHQ-9 is a 9-item patient reported outcome (PRO) used to assess severity of depression. Responses are rated based on the frequency of symptoms on a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day). A PHQ-9 total score ranging from 0 to 27 can be calculated by summing the nine items; a higher score corresponds with more severe depression.
Plasma Concentrations of RO7795081 at Prespecified Timepoints | Predose on Day 1 and at prespecified timepoints until Week 38

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- United States (37):
  - Pinnacle Research Group, Anniston, Alabama
  - Orange County Research Center, Lake Forest, California
  - Prospective Research Innovations Inc., Rancho Cucamonga, California
  - Asclepes Research Centers, Sherman Oaks, California
  - Encompass Clinical Research, Spring Valley, California
  - Chase Medical Research, Waterbury, Connecticut
  - Emerson Clinical Research Institute LLC, Washington D.C., District of Columbia
  - K2 Medical Research-Winter Garden, Clermont, Florida
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research-Maitland, Maitland, Florida
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Accellacare of Duly Health and Care, Oak Lawn, Illinois
  - McFarland Clinic under Accellacare, Ames, Iowa
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Accellacare of Cary, Cary, North Carolina
  - Accellacare - Hickory, Hickory, North Carolina
  - Accellacare of Raleigh, Raleigh, North Carolina
  - Accellacare of Rocky Mount, Rocky Mount, North Carolina
  - Accellacare of Salisbury, Salisbury, North Carolina
  - Accellacare of Piedmont Healthcare, Statesville, North Carolina
  - Accellacare of Wilmington, LLC, Wilmington, North Carolina
  - Accellacare Research of Winston Salem, Winston-Salem, North Carolina
  - Alliance for Multispecialty Research, LLC (AMR Norman), Norman, Oklahoma
  - Tristar Clinical Investigations, Philadelphia, Pennsylvania
  - Internal Medicine and Pediatrics Associates of Bristol, Bristol, Tennessee
  - Alliance for Multispecialty Research. LLC, Knoxville, Tennessee
  - Accellacare of Knoxville, Knoxville, Tennessee
  - Knoxville-Summit-Halls Family Practice, Knoxville, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Apex Mobile Clinical Research, Bellaire, Texas
  - Velocity Clinical Research, Dallas, Texas
  - Juno Research, LLC, Houston, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Manassas Clinical Research Center, Manassas, Virginia

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing